CLINICAL TRIAL: NCT01796561
Title: Effect of Chronic Polyphenol-rich Olive Leaf Extract Intake on Cardiovascular Risk Markers
Brief Title: The Effect of Olive Leaf Extract on Blood Pressure in Overweight Prehypertensives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Massey University (Other)
Responsible Party: Principal Investigator, Jeremy Paul Edward Spencer, Professor of Biochemistry, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OLE chronic study
Record Dates: First submitted 2013-02-20; First posted 2013-02-21 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Olive leaf extract liquid (Active Comparator): 20ml of polyphenol-rich olive leaf extract liquid to be consumed daily for 6 weeks
  Interventions: Dietary Supplement: Olive leaf extract liquid
- Placebo liquid (Placebo Comparator): 20ml of polyphenol-free placebo liquid (containing water, glycerin, flavours, colours and aromas) to be consumed daily for 6 weeks

INTERVENTIONS:
Dietary Supplement: Olive leaf extract liquid — Commercially available polyphenol-rich olive leaf extract liquid
  Arms: Olive leaf extract liquid

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of death in New Zealand (40% of all deaths). 37% of New Zealanders suffer from high blood pressure (World Health Organisation 2008 figures), a well established modifiable risk factor for CVD. Above 115/75 mmHg, CVD risk doubles for each increment of 20/10 mmHg that blood pressure is raised. An increase in BMI and waist circumference has been associated with an increase in blood pressure. The leaves of the olive plant are rich in plant compounds known as polyphenols. This particular group of polyphenols are known secoiridoids, which are also present in olive oil and olives though at lower concentrations, are only found in this family of plants. Diets high in polyphenols have been found to reduce the risk of chronic diseases. Studies have shown that consumption of phenolic-rich olive leaf extract (OLE) can significantly reduce blood pressure in individuals suffering from high blood pressure (hypertension), with the magnitude of effect being comparable to a commonly used antihypertensive drug. In such trials OLE also resulted in an improved blood lipid (a reduction in total and LDL cholesterol and triacylglycerides) which also reduces CVD risk. One study testing the effect of OLE on individuals with mild or prehypertension (i.e. those with systolic blood pressure in the range 121-139 mmHg and diastolic blood pressure in the range 81-89 mmHg but not taking antihypertensive medication) also found these same improvements. OLE has been indicated to have the potential to improve other cardiovascular risk markers such as vascular function, inflammation, platelet aggregation, oxidation of LDL and glucose tolerance however much of this evidence is derived from animal, in vitro and ex vivo studies and so well designed and controlled human studies are required to verify that these findings are applicable to humans. Therefore OLE supplementation may be a useful dietary strategy for reducing CVD risk in a cohort of overweight prehypertensive individuals.

The aim of the study is to determine the effect of OLE intake on blood pressure and other CVD risk markers in overweight subjects with mild hypertension and to link any study outcomes with the presence of OLE phenolics in urine

ELIGIBILITY:
Inclusion Criteria:

Men 18-65 years; Non-smokers; Prepared to consume olive leaf extract liquid Systolic blood pressure 121-139 mmHg and diastolic blood pressure 81-89 mmHg Body mass index (BMI) between 25-30 kg/m2 or waist >102 cm

Exclusion Criteria:

Smokers Using blood pressure, lipid lowering, thyroid disorder, blood clotting medication Using supplements or functional foods that will affect lipid concentrations (e.g. sterol enriched spreads) Chronic disease e.g. CHD, diabetes, cancer, digestive disorders Individuals who are unwilling to refrain from consuming olive containing products for the duration of the study

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Blood pressure measured via 24 hour ambulatory blood pressure monitors | 6 weeks

SECONDARY OUTCOMES:
Vascular function assessed by pulse wave velocity (PWV) | 6 weeks
Lipid profile measured via serum assay | 6 weeks
Inflammatory cytokines measured via plasma assay | 6 weeks
Fructosamine measured via plasma assay | 6 weeks
Glucose measured via plasma assay | 6 weeks
Nitric oxide measured via plasma assay | 6 weeks
Insulin measured via plasma assay | 6 weeks
Haemostatic factors (D-dimer, PAI-1 ag, von Willebrand factor, prothrombin F1+2, factor VIII) measured via plasma assay | 6 weeks
Oxidised LDL measured via plasma assay | 6 weeks
Obesity markers (adiponectin, CCL-2, complement factor D, CRP, IL-6, IL-10, leptin, resistin, serpin E1 and TNF-a) measured via plasma assay | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Welma Stonehouse, PhD, Principal Investigator — Massey University
Locations (1):
- Institute of Food, Nutrition and Human Health, Massey University, Albany, North Shore, Auckland, New Zealand